CLINICAL TRIAL: NCT03984708
Title: New Therapeutic Strategy in ALS Based on Metabolic Status and Associated Metabolic Pathways.
Acronym: METABOCALS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: DR180135; 2019-A00649-48 (Other: IdRCB)
Record Dates: First submitted 2019-06-04; First posted 2019-06-13 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: Amyotrophic Lateral Sclerosis; Metabolomics; Transcriptomics; Biomarkers; Fibroblast
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — Sampling Studies; Calorimetry, Indirect

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Case group (Other): The intervention, specific to the study, is to take samples at baseline on patients with Amyotrophic Lateral Sclerosis
  Interventions: Other: Samples; Other: Indirect calorimetry; Other: Electrical bioimpedance
- Control group (Other): The intervention, specific to the study, is to take samples at baseline on patients without neurological disease
  Interventions: Other: Samples

INTERVENTIONS:
Other: Samples — Blood sample, skin biopsy
Other: Indirect calorimetry — Measurement of energy expenditure by indirect calorimetry
  Arms: Case group
Other: Electrical bioimpedance — Measurement of electrical bioimpedance
  Arms: Case group

SUMMARY:
Amyotrophic lateral sclerosis (ALS) is a neurodegenerative disease that affects central and peripheral motor neurons. None of the clinical trials conducted have been clearly successful and the disease remains incurable, putting patients' vital prognosis at risk in the medium term. An alteration of the basal metabolism leading to hypermetabolism has been described in several articles in the literature. The causes of this hypermetabolism and the precise exploration of the metabolic pathways involved are still poorly understood. The fibroblasts of ALS patients may be the site of some metabolic disturbances in this disease with a hypothetical specific basal metabolic profile. These cells are adapted to different metabolic explorations such as omnic approaches. Superficial skin biopsy followed by fibroblast culture can provide a considerable biobank. This cellular richness will allow us, in ALS patients and their controls, to perform metabolomic and lipidomic approaches, as well as the quantification transcriptomic approach."

DETAILED DESCRIPTION:
Amyotrophic lateral sclerosis (ALS) is a neurodegenerative disease that affects central and peripheral motor neurons. None of the clinical trials conducted have been clearly successful and the disease remains incurable, putting patients' vital prognosis at risk in the medium term. An alteration of the basal metabolism leading to hypermetabolism has been described in several articles in the literature. The causes of this hypermetabolism and the precise exploration of the metabolic pathways involved are still poorly understood. The fibroblasts of ALS patients may be the site of some metabolic disturbances in this disease with a hypothetical specific basal metabolic profile. These cells are adapted to different metabolic explorations such as omnic approaches. Superficial skin biopsy followed by fibroblast culture can provide a considerable biobank. This cellular richness will allow us, in ALS patients and their controls, to perform experiments for the quantification of metabolites by metabolic and lipidomic approaches, as well as the quantification of mRNAs and the rate of gene transcription by a transcriptomic approach.

ELIGIBILITY:
Case group selection criteria:

Inclusion Criteria:

* Age ≥ 18 years and ≥ 75 years
* ALS according to the El Escorial criteria
* Diagnosis of ALS < 6 months
* Symptoms onset < 2 years
* Patients affiliated to social security scheme
* Informed consent signed by the patient

Exclusion Criteria:

* Pregnant or breastfeeding women
* Contraindication to biopsy
* Contraindication to local anesthesia
* Treatment with oral or injectable anticoagulants, antiplatelet (except aspirin)
* Unbalanced Diabetes
* Systemic corticosteroid treatment
* Dermatological diseases of the fibroblast
* Skin cancer
* Protection measure for guardianship or curatorship

Control group selection criteria:

Inclusion Criteria:

* Age ≥ 18 years and ≥ 75 years
* No neuronal disease
* Patients affiliated to social security scheme
* Informed consent signed by the patient

Exclusion Criteria:

* Pregnant or breastfeeding women
* Contraindication to biopsy
* Treatment with oral or injectable anticoagulants, antiplatelet (except aspirin)
* Unbalanced Diabetes
* Systemic corticosteroid treatment
* Dermatological diseases of the fibroblast
* Skin cancer
* Protection measure for guardianship or curatorship

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2020-01-27 (Actual); Primary Completion 2023-01-10 (Actual); Study Completion 2024-03-05 (Actual)

PRIMARY OUTCOMES:
Metabolic signature of fibroblast : concentrations of molecules detected by mass spectrometry | Baseline
  The metabolomic profile of fibroblast represents the combination of the different molecules detected/quantified by mass spectrometry
Metabolic signature of blood : concentrations of molecules detected by mass spectrometry | Baseline
  The metabolomic profile of blood represents the combination of the different molecules detected/quantified by mass spectrometry

SECONDARY OUTCOMES:
Expression levels of targeted molecules using transcriptomics | Baseline
  Choice of molecules based on results obtained by metabolomics approaches

CONTACTS AND LOCATIONS:
Overall Officials: Hélène BLASCO, MD-PhD, Study Director — University Hospital, Tours
Locations (2):
- France (2):
  - Neurology Department, University Hospital, Limoges, Limoges
  - Neurology Department, University Hospitla, Tours, Tours

IPD SHARING:
Plan to Share IPD: No